CLINICAL TRIAL: NCT03905551
Title: The Effect of Exercise Rehabilitation Regimes in Combination With Changes in Dialysis Procedures in Aspects Related to Quality of Life and Health in End Stage Renal Disease Patients
Brief Title: Impact of Cold Dialysis in Combination With Intradialytic Exercise in Aspects Related to Quality of Life and Health
Acronym: REACD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Giorgos K. Sakkas, Professor in Clinical Exercise Physiology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 921-5/11/2014
Record Dates: First submitted 2019-03-29; First posted 2019-04-05 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: cold dialysis; intradialytic exercise; insulin resistance; thermoregulation; muscle architecture; quality of life; fitness; fatigue; physical activity
MeSH Terms: conditions — Insulin Resistance; Fatigue; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The current study is a randomized clinical trial lasting for 7 months. Hemodialysis patients, which fulfilled the inclusion criteria, randomly divided into two groups: a) typical dialysis with dialysate temperature at 37°C (TD+EX) in combination with aerobic intradialytic exercise training, b) cold dialysis with dialysate temperature at 35°C (CD) in combination with aerobic intradialytic exercise training (CD+ET).
  Patients enrolled by a research assistant assigned into the study while the order that the patients assigned to the first scenario was randomly using a computer random number generator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Dialysis (Placebo Comparator): Patients participated in a 7 months exercise trials receiving standard dialysis (at 37oC)
  Interventions: Procedure: Typical Dialysis; Procedure: Exercise
- Cold Dialysis (Experimental): Patients participated in a 7 months exercise trials receiving cold dialysis (at 35oC)
  Interventions: Procedure: Cold Dialysis; Procedure: Exercise

INTERVENTIONS:
Procedure: Cold Dialysis — Dialysate temperature reduced to 35oC for a period of 7 months.
  Arms: Cold Dialysis
Procedure: Typical Dialysis — Dialysate temperature is set at 37oC for a period of 7 months
  Arms: Standard Dialysis
Procedure: Exercise — Aerobic Intradialytic exercise training

SUMMARY:
Despite the tremendous advances in dialysis technology, hemodialysis (HD) is a significant challenge for dialysis patients and quality of their lives[2]. Research has shown for years that dialysate fluid temperature and especially the typical dialysis (TD) temperature at (37°C) are complicated by hemodynamic instability which leading to an increased risk of heat-induced hypotension causing patient discomfort and increased mortality.

Cold dialysis (CD) is defined as the reduction of dialysis fluid temperature to 35-36°C, approximately 1°C below the typical dialysate temperature which ranges between 37-38°C. A number of studies have reported beneficial effects of CD on maintaining hemodynamic stability, minimizes hypotension and exerts a protective effect over major organs including the heart and brain. In addition, current evidence showed the protective effect of CD in cardiac performance during the dialysis session. As the investigators know until today cardiovascular mortality is an important issue for nephrologists that care for ESRD patients, however, many other benefits have been observed on patients' overall health and quality of life levels by used of CD.

The above-mentioned benefits of CD in the hemodynamic stability and the general quality of life of the patients are highlighted even further due to the ever-increasing adoption of intradialytic exercise programs. It has been well established that intradialytic exercise leads to benefits of physiological, functional, and psychological deterioration, which commonly accrues as a consequence of biological aging, catabolic illness, and a sedentary lifestyle, factors that may all contribute to the progressive decline of vitality and quality of life commonly observed in ESRD patients.

However, despite a strong rationale for the implementation of intradialytic exercise programs and the aforementioned benefits of CD, the separate and combined effects of these protocols in aspects related to quality of life and health in ESRD patients have not been investigated to date.

The aim of the current clinical study was to assess the effect of exercise rehabilitation regimes in combination with changes in dialysate temperature in aspects related to quality of life and health in end-stage renal disease patients receiving hemodialysis.

DETAILED DESCRIPTION:
The primary aim of the clinical study was to investigate the combined effect of cold dialysis and aerobic exercise in aspects related to health. More specific:

1. To investigate the thermoregulatory responses of hemodialysis patients under four different hemodialysis protocols.
2. To assess the changes in muscular architecture and functional capacity in dialysis patients after 7 months of intradialytic exercise training.
3. To assess the impact on insulin sensitivity and glucose disposal.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable ESRD patients receiving regular hemodialysis treatment for at least 3 months,
* adequate dialysis delivery Kt/V >1.1
* good compliance of dialysis treatment
* serum albumin >2.5 g/dL
* hemoglobin ≥11g/dL.

Exclusion Criteria:

* Patients with a reason to be in a catabolic state,
* hyperthyroidism,
* active vasculitis,
* malignancies,
* pregnancy
* HIV,
* opportunistic infections,
* musculoskeletal contraindication to exercise,
* requirement for systemic anticoagulation,
* participant or participated in an investigational drug or medical device study within 30 days,
* active inflammations, that required intravenous antibiotics within 3 months prior to enrollment,
* diabetics receiving insulin therapy,
* New York Heart Association grade IV heart failure,
* mental incapacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Body Heat Storage | Changes from baseline at 7 months
  Body Heat storage will be assessed during the 4 hours of dialysis under the two main conditions. Body Heat Storage is calculated in Watt
Change in Insulin Resistance | Changes from baseline at 7 months
  Insulin resistances will be assessed by an Oral Glucose Tolerance Test using the OGIS index
Change in Muscle Size | Changes from baseline at 7 months
  Muscle size will be assessed using Ultrasonography

SECONDARY OUTCOMES:
Change in Quality of life score | Changes from baseline at 7 months
  Quality of life will be assessed using the Sort Form 36 questionnaire. The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is consisted of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The eight sections are:
  * vitality
  * physical functioning
  * bodily pain
  * general health perceptions
  * physical role functioning
  * emotional role functioning
  * social role functioning
  * mental health
Change in Functional Capacity | Changes from baseline at 7 months
  Functional capacity will be assessed by the 6 min walking test
Change in Daily Physical activity | Changes from baseline at 7 months
  Daily physical activity will be assessed by a 7 day recall pedometer

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos K Sakkas, PhD, Principal Investigator — University of Thessaly
Locations (3):
- Greece (3):
  - University Hospital of Larissa, Nephrology Clinic, Larissa, Thessaly
  - Patsidis General Clinic, Larissa, Thessaly
  - General Hospital of Trikala, Trikala, Thessaly

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parnas I, Spira M, Werman R, Bergmann F. Micro-electrode studies of the giant fibres of the American cockroach. Electroencephalogr Clin Neurophysiol. 1969 Aug;27(2):221. No abstract available. PMID 4184202
- [Background] Krase AA, Flouris AD, Karatzaferi C, Giannaki CD, Stefanidis I, Sakkas GK. Separate and combined effects of cold dialysis and intradialytic exercise on the thermoregulatory responses of hemodialysis patients: a randomized-cross-over study. BMC Nephrol. 2020 Dec 2;21(1):524. doi: 10.1186/s12882-020-02167-z. PMID 33267815
- [Derived] Krase AA, Giannaki CD, Flouris AD, Liakos D, Stefanidis I, Karatzaferi C, Sakkas GK. The Acute, Combined, and Separate Effects of Cold Hemodialysis and Intradialytic Exercise in Insulin Sensitivity and Glucose Disposal. ASAIO J. 2024 May 1;70(5):436-441. doi: 10.1097/MAT.0000000000002117. Epub 2024 Jan 23. PMID 38261536
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Krase AA, Terzis G, Giannaki CD, Stasinaki AN, Wilkinson TJ, Smith AC, Zorz C, Karatzaferi C, Stefanidis I, Sakkas GK. Seven months of aerobic intradialytic exercise training can prevent muscle loss in haemodialysis patients: an ultrasonography study. Int Urol Nephrol. 2022 Feb;54(2):447-456. doi: 10.1007/s11255-021-02931-6. Epub 2021 Jun 28. PMID 34184202
- See also: Cold dialysis and its impact on renal patients' health: An evidence-based mini review. — http://www.ncbi.nlm.nih.gov/pubmed/28540201
- See also: The Effect of Cold Dialysis in Motor and Sensory Symptoms of RLS/WED Occurring During Hemodialysis: A Double-Blind Study. — https://www.ncbi.nlm.nih.gov/pubmed/28682991